CLINICAL TRIAL: NCT07294950
Title: Impact of Semaglutide Withdrawal on Cardiometabolic Profile and Physiology of Energy Balance: a Randomized Controlled Trial Comparing Gradual Dose Reduction With Immediate Treatment Cessation.
Brief Title: Impact of Semaglutide Withdrawal on Cardiometabolic Profile and Physiology of Energy Balance: Recovery Effects After Semaglutide Termination
Acronym: REST
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Mount Sinai Hospital, Canada (Other)
Collaborators: Heart and Stroke Foundation of Canada (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REB#1360
Record Dates: First submitted 2025-11-17; First posted 2025-12-19 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2025-10

CONDITIONS: Obesity (Disorder); Weight Change; Blood Pressure Monitoring; Appetite Regulation
Keywords: Randomized controlled trial; Interventional
MeSH Terms: conditions — Obesity; Body Weight Changes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Gradual dose reduction of semaglutide (Experimental): Participants will reduce semaglutide dosage by 25% every 4-weeks until complete treatment cessation at week 16
  Interventions: Drug: Gradual dose reduction of semaglutide
- Cessation of semaglutide (Active Comparator): Participants will discontinue treatment at once at week 16
  Interventions: Drug: Abrupt cessation of semaglutide

INTERVENTIONS:
Drug: Gradual dose reduction of semaglutide — Pparticipants will reduce semaglutide dosage by 25% every 4-weeks until complete treatment cessation at week 16
  Arms: Gradual dose reduction of semaglutide
Drug: Abrupt cessation of semaglutide — Cessation of semaglutide at 16-weeks
  Arms: Cessation of semaglutide

SUMMARY:
Semaglutide is a medication from the class of drugs called glucagon-like peptide-1 agonists that promote weight loss. There is little clinical data on the best strategy to achieve weight maintenance following weight reduction induced by semaglutide. For people who need to discontinue treatment, it is unknown whether the weight regain, its accompanied health benefits could be ameliorated with a gradual reduction in semaglutide. The investigators will study if a gradual reduction of semaglutide is associated with different heart risk profile and hormones involved in energy regulation as compared to immediate treatment cessation.

DETAILED DESCRIPTION:
It is known that semaglutide induces a supra-physiologic agonism of GLP-1 receptors on central nervous system receptors associated with hedonic eating which likely promotes a homeostatic response (i.e. adaptation) related to appetite control. This concept raises the question of whether a gradual de-escalation of GLP-1RA could ameliorate the tendency for weight regain/cardiometabolic deterioration and compensatory changes in energy balance regulation following cessation of treatment.Thus, the investigators propose an open-label, parallel-arm, randomized controlled trial to determine whether a gradual dose reduction in semaglutide prior to complete discontinuation is associated with differential changes in weight and cardiometabolic profile (blood pressure homeostasis and energy balance regulatory hormones) as compared to immediate treatment cessation in individuals living with obesity without pre-existing cardiovascular disease who are receiving semaglutide for weight management.

ELIGIBILITY:
Inclusion Criteria:

* Men and women with previously diagnosed BMI ≥ 30 kg/m2 or BMI ≥ 27 kg/m2 and adiposity-related complications (such as osteoarthritis, nonalcoholic liver disease, sleep apnea, and hypertension) without preexisting cardiovascular disease or type 2 diabetes.
* Age 18 - 75 years inclusive
* Ongoing weight-loss treatment consisting of weekly subcutaneous semaglutide at minimum dose of 1 mg/weekly with documented weight reduction of at least 10% of pre-treatment body weight
* Stable weight over past 12 weeks (less than 5% change in body weight) (self-reported)
* Ability to read and understand English

Exclusion Criteria:

* Previously diagnosed cardiovascular disease defined as previous myocardial infarction, previous stroke, or symptomatic peripheral arterial disease.
* Currently pregnant or lactating
* Previously diagnosed type 2 diabetes
* Use of any other pharmacological treatment for weight-loss
* Previous surgical treatment for weight loss such as gastric bypass or gastric band
* Any history of eating disorder
* Renal dysfunction as evidenced by estimated glomerular filtration rate < 25 ml/min by CKD-EPI Creatinine Equation
* New York Heart Association class II-IV heart failure
* Hepatic disease considered to be clinically significant (includes jaundice, chronic hepatitis, or previous liver transplant) or transaminases >2.5X the upper limit of normal
* Malignant neoplasm requiring chemotherapy, surgery, radiation or palliative therapy within the previous 5 years (with the exception of basal cell skin cancer)
* Personal or family history of medullary thyroid carcinoma or in patients with Multiple Endocrine Neoplasia syndrome type 2
* Any other factor likely to limit adherence to the study, in the opinion of the investigators

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Estimated)
Dates: Start 2026-02-01 (Actual); Primary Completion 2028-09 (Estimated); Study Completion 2029-05 (Estimated)

PRIMARY OUTCOMES:
Differences in changes in body weight between each study group | 32 weeks
  Differences in body weight change (%) between baseline visit 1 (semaglutide discontinuation) and 5 (16-weeks after complete semaglutide withdrawal) will be compared between the study groups

SECONDARY OUTCOMES:
Differences in 24-h systolic BP levels between each study group | 32 weeks
  Systolic BP will be assessed as the difference in 24-h ambulatory systolic BP between the study groups at visit 5 (16-weeks after complete semaglutide withdrawal)
Differences in fasting ghrelin between each study group | 32 weeks
  Differences in fasting ghrelin between the study groups will be assessed at week 5 (16-weeks after complete semaglutide withdrawal)

OTHER OUTCOMES:
Changes in body mass index (BMI) | 32 weeks
  Changes in BMI [calculated as weight / height2 (in kg/m2)] between baseline visit 1 (semaglutide discontinuation) and 5 (16-weeks after complete semaglutide withdrawal) will be compared between the study groups
Changes in waist circumference | 32 weeks
  Changes in waist circumference between baseline visit 1 (semaglutide discontinuation) and 5 (16-weeks after complete semaglutide withdrawal) will be compared between the study groups

CONTACTS AND LOCATIONS:
Locations (1):
- Leadership Sinai Centre for Diabetes, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No